CLINICAL TRIAL: NCT00425685
Title: Use of Extracorporeal Membrane Oxygenation in Treatment of Acute Myocardial Infarction Following Cardiac Surgery Procedures
Brief Title: Use of ECMO in Acute MI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Other Study IDs: Use of ECM in acute MI; ECMO and AMI
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2007-01-23 (Estimated); Status verified 2007-01

CONDITIONS: ECMO and Acute MI
Keywords: cardiopulmonary resuscitation, ECMO, shock, survival, heart failure, transplantation, heart assist device.
MeSH Terms: conditions — Shock; Heart Failure

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
ECMO offers an acceptable cardiopulmonary support in adults with similar hospital survival rates as other mechanical support. It is versatile and salvages some patients, who may otherwise die. Improvement in intermediate term outcome will require multidisciplinary approach to protect organ function and limit organ injury during this support.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is an established treatment option in patients with Cardiogenic Schock. We retrospectively reviewed early and mid-term outcome as well as predictors of survival during using ECMO. This report reviews our experience with this support system in last 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Acute MI

Exclusion Criteria:

* Contraindication against ECMO

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-01; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Bakhtiary, MD, Principal Investigator — JW Goethe University